CLINICAL TRIAL: NCT06239948
Title: The Brain Symphony For Post-Stroke Rehabilitation - A Pilot Randomized Controlled Study With P.Ramlee Songs
Brief Title: The Brain Symphony For Post-Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Brain Symphony
Record Dates: First submitted 2024-01-16; First posted 2024-02-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2024-01

CONDITIONS: Stroke
Keywords: Music Listening; Stroke; Rehabilitation; Transcranial Magnetic Stimulation (TMS); Neuroplasticity; P. Ramlee Music
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The participants were categorized into two groups: stroke survivors and healthy individuals and randomized into control group (without music) and experimental group (with music).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): without music
  Interventions: Other: Without Music
- experimental group (Experimental): with music
  Interventions: Other: With Music

INTERVENTIONS:
Other: With Music — each subject was placed in a TMS laboratory with music for 20 minutes
  Arms: experimental group
Other: Without Music — each subject was placed in a TMS laboratory without music for 20 minutes
  Arms: control group

SUMMARY:
Music listening intervention has made great strides in improving the condition of stroke survivors. Thus, this research explores the effects of music listening intervention on post-stroke survivors during rehabilitation by using P. Ramlee songs.

DETAILED DESCRIPTION:
Objective: Music listening intervention has made great strides in improving the condition of stroke survivors. Thus, this research explores the effects of music listening intervention on post-stroke survivors during rehabilitation by using P. Ramlee songs.

Materials & Methods: In the first phase, surveys were conducted to determine the selection of songs to be used in the second phase. The second phase is applying music listening intervention on a small sample of 20 subjects, aged 55 years old and above. The participants were categorized into two groups: stroke survivors and healthy individuals and randomized into control group (without music) and experimental group (with music). The second phase consists of three stages. Stage one is to pre-screen and select potential subjects before the experiment. The second stage aims to determine the effect of P. Ramlee music on stroke survivors during their rehabilitation through augmenting their brain neuroplasticity with measurement of the MEP using TMS. The final stage compares the effects of MEP between lesion and non-lesion areas.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No history of seizures or epilepsy
* Able to hear well
* Able to attend experiment sessions without scheduling conflicts
* No contraindications to undergoing TMS

Exclusion Criteria:

• None

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Transcranial Magnetic Stimulation (TMS) | 24 months
  Wilcoxon signed-ranks test for the comparison of pre- and post- experiment

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No